CLINICAL TRIAL: NCT05262322
Title: A Descriptive Non-interventional Study to Evaluate the Use of Direct Oral Anticoagulants in UK Clinical Practice for Patients With a First Stroke Attributable to Nonvalvular Atrial Fibrillation
Brief Title: Study to Evaluate the Use of Direct Oral Anticoagulants in UK Clinical Practice For Patients With a First Stroke Attributable to Nonvalvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo UK Ltd, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: EDX/18/0414(2)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Direct oral anticoagulants; Edoxaban; Apixaban; Rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; apixaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All Participants (Group 1; Retrospective): All participants' data will be collected retrospectively from medical records 12 months prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
- Subset of All Participants (Group 2; Prospective): A subset of participants from Group 1 who were initiated on apixaban, edoxaban or rivaroxaban for secondary prophylaxis of stroke will take part in this prospective component of the study, whereby data on their management pathway (treatments and follow-up appointments) and patient-reported outcomes will be collected for 6 months from the date of first dose of DOAC treatment.
  Interventions: Drug: Edoxaban; Drug: Apixaban; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Edoxaban — This was a non-interventional, observational study. No drug was administered in this study.
  Groups: Subset of All Participants (Group 2; Prospective)
Drug: Apixaban — This was a non-interventional, observational study. No drug was administered in this study.
  Groups: Subset of All Participants (Group 2; Prospective)
Drug: Rivaroxaban — This was a non-interventional, observational study. No drug was administered in this study.
  Groups: Subset of All Participants (Group 2; Prospective)

SUMMARY:
National Institute of Health and Care Excellence (NICE) guidance recommends anticoagulation for stroke prevention in high risk patients with nonvalvular atrial fibrillation (AF).

Early evidence suggest that patients with atrial fibrillation (AF) who do not receive anticoagulation are more likely to experience a stroke. However, the characteristics of patients experiencing a first AF-related stroke in real-world settings, who have not been receiving anticoagulation, have not been well documented.

It is unclear how the direct anti-FXa oral anticoagulants have been used within real world practice since the introduction of edoxaban in 2015.

DETAILED DESCRIPTION:
This non-interventional study will focus specifically on the patient characteristics, management pathways, and patient reported experiences associated with real world use of three direct anti-FXa oral anticoagulants (DOAC) commonly used within United Kingdom clinical practice; apixaban, rivaroxaban and edoxaban.

The primary objective will describe the demographics, clinical characteristics and medical history of patients presenting with a first ischaemic stroke with AF who have not received anticoagulation (for any reason) in the 12 months prior to stroke, by type of anticoagulant treatment subsequently prescribed for secondary prophylaxis of stroke.

Secondary objectives of the study will describe management pathways of patients initiated on DOACs (apixaban, edoxaban or rivaroxaban) for secondary prophylaxis of stroke, including timing and reasons for any dose changes or treatment switches to alternative anticoagulants; describe hospital resource use and clinical assessments associated with DOAC treatment for secondary prophylaxis of stroke; describe real world patient-reported adherence to DOACs for secondary prophylaxis of stroke; and describe patient experience and treatment satisfaction for patients receiving DOAC therapy for secondary prophylaxis of stroke.

ELIGIBILITY:
Inclusion Criteria:

- For all patients:

* Participants presenting to the study centre with a first ischaemic stroke which is, in the clinician's opinion, attributable to nonvalvular AF
* Participants aged 18 years or over at time of first stroke

For group 2 patients:

* Participants initiated on apixaban, edoxaban or rivaroxaban after their first stroke

Exclusion Criteria:

* For all patients:

  * Participants prescribed any anticoagulant for any purpose in the 12 months prior to stroke diagnosis
  * Participants with haemorrhagic stroke
  * Participants with diagnosis of transient ischemic attack
  * Participants with severe cognitive or emotive deficit
  * Participants whose medical records are not available for review
  * Participant unwilling or unable to give written informed consent
* For group 2 patients:

  * Participant unwilling or unable to complete the patient-reported questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the wider retrospective study (Group 1 patients), potentially eligible participants will be identified by members of the direct care team from local department databases. Eligible participants will be selected in consecutive chronological order by the direct care team according to the date of stroke diagnosis until the required sample size or the center-specific recruitment target is reached, over a one-year recruitment period.
  The first 50 eligible and consenting participants initiated on either apixaban, edoxaban or rivaroxaban at any of the study centers during the 28 month recruitment period will also be included in the prospective component of the study.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Mean CHA2DS2-VASc Risk Scores In Participants Presenting With A First Stroke with Atrial Fibrillation (AF) Who Have Not Received Anticoagulation Within 12 Months Prior to Stroke | 12 month period prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
  CHA2DS2-VASc risk scores range from 0-9, where a score of 0 is "low" risk of stroke, 1 is "moderate", and any score above 1 is a "high" risk. Scores will be calculated based on relevant demographic and clinical data recorded in medical notes for pre-index observation period.

SECONDARY OUTCOMES:
Mean Time from Atrial Fibrillation (AF) Diagnosis Until Stroke In Participants Presenting With A First Stroke with Atrial Fibrillation Who Have Not Received Anticoagulation Within 12 Months Prior to Stroke | Approximately 12 month period prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
  The time from AF diagnosis until stroke will be assessed.
Stroke Severity In Participants Presenting With A First Stroke with Atrial Fibrillation (AF) Who Have Not Received Anticoagulation Within 12 Months Prior to Stroke | Approximately 12 month period prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
  Stroke severity will be assessed by NIHSS classification (mild, moderate, moderate to severe, and severe), Oxfordshire Community Stroke Project Score, classification based on CT scan, and opinion of treating clinician.
Number of Participants With Relevant Cardiovascular and Related Non-Cardiovascular Conditions In Participants Presenting With A First Stroke with Atrial Fibrillation Who Have Not Received Anticoagulation Within 12 Months Prior to Stroke | Approximately 12 month period prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
  Cardiovascular and related non-cardiovascular events, such as hypertension, congestive heart failure, vascular disease (peripheral artery disease, previous myocardial infarction, aortic plaque), diabetes mellitus, renal impairment, renal failure, hepatic failure, coronary artery disease, carotid artery disease, reduced ejection fraction, liver disease, and other, will be assessed.
Number of Participants Receiving Concomitant Medications At Time of First Stroke and Newly Prescribed Within 1 Month After Stroke | Approximately 12 month period prior to the date of diagnosis of a first ischaemic stroke attributable to nonvalvular AF
  Concomitant medications may include: beta blockers, diuretics, antiplatelet agents (e.g. aspirin), ACE (angiotensin-converting-enzyme) inhibitors, ATII-receptor antagonists, statins, ASA (acetylsalicylic acid), and P-gp (P-glycoprotein) inhibitors.
Type of First Anticoagulant Medication Prescribed After Stroke In Participants Presenting With A First Stroke with Atrial Fibrillation Who Have Not Received Anticoagulation Within 12 Months Prior to Stroke | Within 1 month after stroke
  Anticoagulant medications may include apixaban, edoxaban, rivaroxaban, warfarin, dabigatran, and other.
Time From Stroke to First Dose of Direct Oral Anticoagulant (DOAC) in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | From stroke to first dose of DOAC, up to 6 months after date of first dose of DOAC
  The time from stroke to first dose of anticoagulant medication will be assessed.
Time to Discontinuation of First Direct Oral Anticoagulant (DOAC) Treatment in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Up to 6 months after date of first dose of DOAC
  The time to discontinuation of anticoagulant medication will be assessed.
Number of Participants Receiving Clinical Assessments in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Up to 6 months after date of first dose of DOAC
  Clinical assessments may include weight, coagulation screens (international normalized ratio), full blood count (FBC), urea and electrolyte tests (U&E), renal function and liver function tests (alanine transaminase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], albumin and bilirubin tests) as well as other neurological, heart or functional assessments (thyroid function tests, blood pressure, 12 lead ECG/EKG including heart rate, echocardiography and relevant imaging CT scan, ultrasound, MRI and PET scans.
Number of Secondary Care Visits in 6 Months Post-first Direct Oral Anticoagulant (DOAC) Dose in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Up to 6 months after date of first dose of DOAC
  Secondary visits will include inpatient, outpatient, and accident and emergency.
Duration of Inpatient Stays in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Up to 6 months after date of first dose of DOAC
  The length of inpatient hospital stays will be assessed.
Mean Absolute Morisky Medication Adherence Scale (MMAS-8) Score After First Direct Oral Anticoagulant (DOAC) Dose in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Up to 6 months after date of first dose of DOAC
  Morisky Medication Adherence Scale (MMAS-8) range from 0 to 8, where higher scores indicate medication adherence and lower scores indicate nonadherence. Medication adherence will be assessed at 3 and 6 months.
Number of Participants Taking Direct Oral Anticoagulant (DOAC) Medication Within Past 7 Days in Participants Who Are Initiated on Apixaban, Edoxaban, or Rivaroxaban | Within past 7 days
  Anticoagulant medication may include apixaban, edoxaban, rivaroxaban, warfarin, dabigatran, and other. DOAC medication will be assessed at 3 and 6 months.
Mean Absolute Treatment Satisfaction Questionnaire for Medication (TSQM) Score Post-first Direct Oral Anticoagulant Dose | Up to 6 months after date of first dose of DOAC
  Treatment Satisfaction Questionnaire for Medication (TSQM) domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain. Treatment satisfaction will be assessed at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde, Glasgow
  - Gloucestershire Royal Hospital - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - Leicester Royal Infirmary - University Hospitals of Leicester NHS Trust, Leicester
  - St George's Hospital - St George's University Hospital's NHS Foundation Trust, London
  - Royal Victoria Infirmary - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Royal Gwent Hospital - Aneurin Beban University Health Board, Newport
  - Musgrove park Hospital - Taunton and Somerset NHS Foundation Trust, Taunton
  - Yeovil District Hospital - Yeovil District Hospital NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: No